CLINICAL TRIAL: NCT04177719
Title: Understanding the Neurobiological Effects of Oxytocin on Social Trust Deficits in Schizophrenia: A Multimodal Imaging - Genetics Study
Brief Title: Neurobiological Effects of Oxytocin in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dr Naren P Rao, Additional Professor of Psychiatry, National Institute of Mental Health and Neuro Sciences, India
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 00908
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Single-dose oxytocin or placebo will be given intranasally on separate scan days. The order of administration will be counterbalanced
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Single-dose oxytocin or placebo will be given intranasally on separate scan days. The order of administration will be counterbalanced
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — oxytocin will be given intranasally. The order of administration will be counterbalanced
  Arms: Oxytocin
Drug: Placebo — Saline placebo will be given intranasally. The order of administration will be counterbalanced
  Arms: Placebo

SUMMARY:
22 male patients with schizophrenia and 22 male healthy volunteers will be included in the study. Subjects who meet the inclusion and exclusion criteria for the study will be recruited. After completion of clinical assessments and neuropsychological assessments, all subjects will undergo two multi-modal imaging sessions. In one scan they will receive intranasal oxytocin and in another scan will receive intranasal saline as control. The order of administration of the medication will be counterbalanced and subjects will be blind to the medication administered. Using the simultaneous PET-MRI scanner, PET and fMRI data will be collected simultaneously. Blood will be collected for analysis of oxytocin receptor gene polymorphism and its potential effect on brain activity.

ELIGIBILITY:
Schizophrenia group

Inclusion Criteria:

1. Diagnosis of schizophrenia or schizoaffective disorder
2. Males between 18 and 45 years
3. capacity to provide informed consent

Exclusion Criteria:

1. current comorbid axis I diagnosis and no alcohol/substance abuse/dependence in the last 12 months (except nicotine)
2. Contraindication to oxytocin like hypersensitivity, vascular disease, chronic nephritis, epilepsy, asthma
3. Contraindication to MRI like implants/claustrophobia
4. Past history of head injury resulting in loss of consciousness or neurosurgery
5. Concomitant severe medical conditions
6. On treatment with benzodiazepine medications for at least 8 weeks
7. Contraindication to Positron emission tomography

Healthy volunteers

Inclusion Criteria:

1. Males between 18 and 45 years
2. capacity to provide informed consent

Exclusion Criteria:

1. Lifetime diagnosis of psychiatric illness including substance dependence
2. contraindication to oxytocin like hypersensitivity, vascular disease, chronic nephritis, epilepsy, asthma
3. contraindication to MRI like implants/claustrophobia
4. past history of head injury resulting in loss of consciousness or neurosurgery
5. concomitant severe medical conditions
6. on treatment with benzodiazepine medications for at least 8 weeks
7. contraindication to Positron emission tomography
8. Family history of schizophrenia, schizoaffective or schizophreniform disorder in family member

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
PET | 90 minues
  changes in [18F] flumazenil specific binding
fMRI changes | 90 minutes
  changes in brain functional connectivity
MRS | 90 minutes
  Changes in brain chemistry measured using MRS

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health and Neurosciecnes, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No